CLINICAL TRIAL: NCT04884581
Title: The CHANGE Study: Characterization Helping the Assessment of Colorectal Neoplasia in Gastrointestinal Endoscopy
Brief Title: Characterization of Colorectal Neoplasia
Acronym: CHANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuovo Regina Margherita Hospital (Other)
Responsible Party: Principal Investigator, Cesare Hassan, MD, Nuovo Regina Margherita Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHANGE Study
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GI Genius CADx device (Experimental)
  Interventions: Device: GI Genius CADx device

INTERVENTIONS:
Device: GI Genius CADx device — GI Genius System is an Intelligent Endoscopy Module designed to be an adjunct to video colonoscopy with the purpose of supporting the operating physician with artificial intelligence during colonoscopy. GI Genius CADx is the AI software that provides a histology prediction of framed polyps during real-time colonoscopy, with each polyp being classified as adenoma or non-adenoma.

SUMMARY:
This is a post-marketing, single-arm, prospective study investigating the use of GI Genius CADx device in the real-time characterization of colorectal polyps (i.e. prediction of their histology during the colonoscopy). Patients enrolled will undergo a standard white-light colonoscopy with the support of the latest version of the CE-marked GI Genius CADx device. Colonoscopy will be performed according to the standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years or older undergoing screening colonoscopy for CRC
* Ability to provide written, informed consent (approved by EC) and understand the responsibilities of trial participation

Exclusion Criteria:

* subjects at high risk for colorectal cancer
* subjects with a personal history of CRC, IBD or hereditary polyposis or non-polyposis syndromes
* patients with previous resection of the sigmoid rectum
* patients on anticoagulant therapy, which precludes resection / removal operations due to histopathological findings
* patients who perform an emergency colonoscopy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Negative Predictive Value (NPV) | 4 months
  Negative Predictive Value (NPV) of GI Genius CADx optical diagnosis on diminutive (≤5 mm) rectosigmoid polyps

OTHER OUTCOMES:
Post-polypectomy surveillance interval | 4 months
  Agreement in assignment of post-polypectomy surveillance intervals of the enrolled patients according to established guidelines between the combined use of GI Genius CADx as optical diagnosis for diminutive (≤5 mm) polyps and conventional histology as diagnostic tool for polyps > 5 mm, and histology as diagnostic tool for all the resected polyps (regardless of size or location)
Performance metrics of GI Genius CADx | 4 months
  Sensitivity, Specificity, Accuracy, PPV and NPV of GI Genius CADx optical diagnosis
Performance metrics of the endoscopist with the aid of GI Genius CADx | 4 months
  Sensitivity, Specificity, Accuracy, PPV and NPV of the optical diagnosis of endoscopists assessing lesions in white-light with the help of GI Genius CADx.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuovo Regina Margherita, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brenner TA, Labaki C, Feuerstein JD, Berzin TM. Prospective Validation of the First US FDA-Approved Computer-Aided Quality Assessment Tool for Colonoscopy: An Initial Clinical Experience. Am J Gastroenterol. 2025 Nov 19. doi: 10.14309/ajg.0000000000003855. Online ahead of print. PMID 41257531
- [Derived] Hassan C, Balsamo G, Lorenzetti R, Zullo A, Antonelli G. Artificial Intelligence Allows Leaving-In-Situ Colorectal Polyps. Clin Gastroenterol Hepatol. 2022 Nov;20(11):2505-2513.e4. doi: 10.1016/j.cgh.2022.04.045. Epub 2022 Jul 11. PMID 35835342